CLINICAL TRIAL: NCT02554474
Title: Effective of Online Physical Activity Monitoring in Inflammatory Arthritis (OPAM-IA): A New Model of Care
Brief Title: OPAM-IA: Using Digital Activity Trackers to Improve Physical Activity in Inflammatory Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Simon Fraser University (Other); Arthritis Research Centre of Canada (Other); Vancouver General Hospital (Other); The Arthritis Society, Canada (Other); Fraser Health (Other)
Responsible Party: Principal Investigator, Linda Li, Professor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: H15-01843
Record Dates: First submitted 2015-09-16; First posted 2015-09-18 (Estimated); Results first posted 2021-06-04 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Joint Diseases; Rheumatoid Arthritis; Systemic Lupus Erythematosus
Keywords: Physical activity; Exercise; Rheumatoid; Arthritis; Lupus; SLE
MeSH Terms: conditions — Joint Diseases; Arthritis, Rheumatoid; Lupus Erythematosus, Systemic; Motor Activity; Arthritis | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Group (Active Comparator): Time spent in Moderate/Vigorous Physical Activity (MVPA) was measured with a SenseWear Mini sensor over a 7-day period. The mean time was calculated in bouted MVPA per day. A bout is defined as >= 10 consecutive minutes or more at the level of >= 3 METs (i.e., the lower bound of MVPA), with allowance for interruption of up to two minutes below the threshold.
  Interventions: Behavioral: Education, Fitbit/FitViz, physiotherapist counselling.
- Delay Group (Placebo Comparator): Time spent in sedentary activity was measured with a SenseWear Mini sensor over a 7-day period. The mean daily time spent in sedentary activity was calculated with an energy expenditure of <=1.5 METs, occurring in bouts of >= 20 minutes during waking hours.
  Interventions: Behavioral: Same intervention with a 9-week delay

INTERVENTIONS:
Behavioral: Education, Fitbit/FitViz, physiotherapist counselling. — Participants will receive a brief education session, use a physical activity tracker Fitbit Flex with paired with a FitViz app, and remote counseling by a PT. Intervention will be received immediately.
  Arms: Immediate Group
Behavioral: Same intervention with a 9-week delay — The Delayed Intervention Group will receive the same intervention as the Immediate Intervention Group, but with a 9-week delay.
  Arms: Delay Group

SUMMARY:
Being physically active can reduce pain and fatigue, improve mobility and enhance quality of life in people with arthritis, but adherence to an active lifestyle is poor, with less than half of people with arthritis being active. The primary goal of this randomized controlled trial is to assess the efficacy of a physical activity coaching model to improve physical activity participation and reduce sedentary time in patients with Rheumatoid Arthritis and Systemic Lupus Erythematosus. This model combines the use of a Fitbit Flex (wireless physical activity tracker) paired with a FitViz application, a group education session, and telephone counselling by a physiotherapist.

DETAILED DESCRIPTION:
Patient self-management is a fundamental component in arthritis care that is often neglected. Physical activity is an essential part of self-management, however, less than half of people with arthritis are active. There are several factors that are associated with low physical activity participation such as motivation, doubts about the effectiveness of prescribed exercises, and lack of health professional advice on ways to progress physical activity. The variety of risk factors highlights the need for a multifaceted approach that provides support in terms of knowledge, skill development and timely advice from health professionals, as well as motivational support to stay active.

Our primary objective is to assess the efficacy of a physical activity counselling model, involving the use of a Fitbit Flex (wireless physical activity tracker) paired with a FitViz application (app), a group education session, and telephone counselling by a physiotherapist, to improve physical activity participation in patients with rheumatoid arthritis (RA) and systemic lupus erythematosus (SLE). Our secondary objective is to assess the effect of the intervention on reducing patients' sedentary time, and improving fatigue, mood, pain, and self-efficacy in arthritis management. We will carry out three aims: 1) To develop the FitViz app to pair with Fitbit to enhance user experience, 2) To conduct a pilot test for the Fitbit/FitViz intervention, 3) To evaluate the effect of the physical activity coaching model in patients with RA and SLE. In this proof-of-concept randomized controlled trial (RCT), the investigators hypothesize that compared to a control group (i.e. the Delayed Intervention group), participants in the Immediate Intervention Group will 1) increase moderate/vigorous physical activity (MVPA), 2) reduce sedentary time, 3) improve in fatigue, mood, and pain levels, and 4) improve in their self-efficacy in disease management.

The investigators will use a mixed-methods approach, involving a RCT and in-depth interviews. The proof-of-concept study will employ a stepped wedge RCT design, whereby the intervention will be sequentially rolled out to participants over a number of time periods. The order in which individuals receive the intervention will be determined at random. The strength of this design is that it can properly address the efficacy question, while avoiding the dilemma of withholding the intervention to some participants, as in a parallel group design.

ELIGIBILITY:
Inclusion Criteria:

* Have a physician confirmed diagnosis of RA or SLE.
* Have an email address and daily access to a computer with internet connection.
* Be able to attend a 1.5-hour education session at Mary Pack Arthritis Centre, Arthritis Research Centre, or a Fraser Health site.

Exclusion Criteria:

* Have previously used any physical activity wearables.
* Face a level of risk by exercising as identified by the Physical Activity Readiness Questionnaire (PAR-Q).

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-08-25 (Actual); Study Completion 2019-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Li, PhD, Principal Investigator — Professor
Locations (1):
- Arthritis Research Canada, Richmond, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li LC, Feehan LM, Shaw C, Xie H, Sayre EC, Avina-Zubeita A, Grewal N, Townsend AF, Gromala D, Noonan G, Backman CL. A technology-enabled Counselling program versus a delayed treatment control to support physical activity participation in people with inflammatory arthritis: study protocol for the OPAM-IA randomized controlled trial. BMC Rheumatol. 2017 Nov 28;1:6. doi: 10.1186/s41927-017-0005-4. eCollection 2017. PMID 30886950
- [Result] Li LC, Feehan LM, Xie H, Lu N, Shaw C, Gromala D, Avina-Zubieta JA, Koehn C, Hoens AM, English K, Tam J, Therrien S, Townsend AF, Noonan G, Backman CL. Efficacy of a Physical Activity Counseling Program With Use of a Wearable Tracker in People With Inflammatory Arthritis: A Randomized Controlled Trial. Arthritis Care Res (Hoboken). 2020 Dec;72(12):1755-1765. doi: 10.1002/acr.24199. PMID 32248626
- [Result] Leese J, Zhu S, Townsend AF, Backman CL, Nimmon L, Li LC. Ethical issues experienced by persons with rheumatoid arthritis in a wearable-enabled physical activity intervention study. Health Expect. 2022 Aug;25(4):1418-1431. doi: 10.1111/hex.13481. Epub 2022 Mar 18. PMID 35303379
- [Derived] Feehan L, Xie H, Lu N, Li LC. Twenty-four hour physical activity, sedentary behaviour and sleep profiles in adults living with rheumatoid arthritis: a cross-sectional latent class analysis. J Act Sedentary Sleep Behav. 2024 Apr 17;3(1):10. doi: 10.1186/s44167-024-00049-5. PMID 40217417

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period was 2017-2019. Participants were recruited from the Mary Pack Arthritis Program (Vancouver Coastal Health Authority) and Fraser Health Authority in British Columbia, Canada. Study information was also posted on Facebook, Twitter, Kajiji and Craigslist.
Pre-assignment Details: After completing baseline measures at home, participants were randomized to the Immediate or Delay Group in 1:1 allocation ratio.
Groups:
- Immediate Group: Education, Fitbit/FitViz, physiotherapist counselling. These 3 components will be delivered to the participants in Months 1 and 2. The session will include a short presentation about physical activity in everyday life, an individual goal-setting session with a registered PT, and an orientation to the Fitbit and FitViz app. Participants will use the Fitbit/FitViz. The PT will review the progress with participants via bi-weekly phone calls and progressively modify their activities. In Month 3-6, participants will continue using the Fitbit/FitViz and have access to a PT via email as needed, but no bi-weekly phone calls.
  Education, Fitbit/FitViz, physiotherapist counselling.: Participants will receive a brief education session, use a physical activity tracker Fitbit Flex with paired with a FitViz app, and remote counseling by a PT. Intervention will be received immediately.
- Delay Group: Same intervention with a 2 month delay: The full intervention will be initiated in Month 3 and 4 with a brief education session, use of a Fitbit paired with the FitViz app, and counseling by a PT. In Month 5-6, participants will continue the intervention without the PT phone calls, but will have email access to PT, if needed.
  Same intervention with a 2 month delay: The Delayed Intervention Group will receive the same intervention as the Immediate Intervention Group, but with a 2 month delay.
Period: Overall Study
Arm/Group | Immediate Group | Delay Group
Started | 59 | 59
Completed | 56 (Indicates number of participants who completed assessment at the primary endpoint.) | 57 (Indicates number of participants who completed assessment at the primary endpoint.)
Not Completed | 3 | 2
Not completed — Protocol Violation | 1 | 1
Not completed — Health issue not related to the study | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Immediate Group: Education, Fitbit/FitViz, physiotherapist counselling. These 3 components were delivered to the participants in Weeks 1-8. The session included a short presentation about physical activity in everyday life, an individual goal-setting session with a registered PT, and an orientation to the Fitbit and FitViz app. Participants used a Fitbit and the FitViz app. The PT reviewed the progress with participants via bi-weekly counselling phone calls and progressively modify their activities. In Weeks 9-26, participants continued using the Fitbit and FitViz and had access to a PT via email as needed, but no bi-weekly phone calls.
- Delay Group: Same intervention (Education, Fitbit/FitViz, physiotherapist counselling) with a 9-week delay. The full intervention was delivered in Week 10-17. In Weeks 18-26, participants continued using the Fitbit and FitViz and had access to a PT via email as needed, but no bi-weekly phone calls.
- Total: Total of all reporting groups
Arm/Group | Immediate Group | Delay Group | Total
Number analyzed (Participants) | 59 | 59 | 118
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.5 (14.7) | 53.1 (12.6) | 53.3 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 54 | 105
  Male | 8 | 5 | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Daily time in moderate/vigorous physical activity [Mean (Standard Deviation); unit: Minutes] | 37.8 (39.6) | 31.6 (42.7) | 34.7 (41.1)
Time in purposeful activity [Mean (Standard Deviation); unit: Minutes] | 13.0 (20.4) | 11.2 (24.5) | 12.1 (22.5)
Daily steps [Mean (Standard Deviation); unit: Steps] | 5900.8 (3214.1) | 5605.7 (2865.1) | 5753.2 (3035.2)
Daily sedentary time [Mean (Standard Deviation); unit: Minutes] | 491.6 (192.5) | 523.0 (194.4) | 507.3 (193.3)
McGill Pain Questionnaire [Mean (Standard Deviation); unit: Units on a scale] — McGill Pain Questionnaire (range 0-45; lower score = less severe pain)
  Units on a scale | 13.3 (10.8) | 13.9 (9.5) | 13.6 (10.1)
Fatigue Severity Scale [Mean (Standard Deviation); unit: Units on a scale] — Fatigue Severity Scale (range 1-7; lower score = less fatigue)
  Units on a scale | 4.8 (1.4) | 4.9 (1.3) | 4.8 (1.3)
Partners in Health [Mean (Standard Deviation); unit: Units on a scale] — Partners in Health (range 0-96; higher score = higher perceived confidence and ability in self-care)
  Units on a scale | 72.8 (11.7) | 73.5 (12.2) | 73.1 (11.9)
Patient Health Questionnaire (PHQ-9) [Mean (Standard Deviation); unit: Units on a scale] — PHQ-9; range 0-27; lower score = less depressive symptoms
  Units on a scale | 7.6 (5.9) | 8.1 (5.6) | 7.8 (5.7)
Self-Reported Habit Index [Mean (Standard Deviation); unit: units on a scale] — Sitting at work subscale, Sitting at Leisure subscale, Walking subscale (range 1-7; higher score = stronger habit)
  units on a scale
    Sitting at work subscale | 4.5 (1.7) | 4.6 (1.8) | 4.5 (1.7)
    Sitting at leisure subscale | 4.7 (1.4) | 4.7 (1.3) | 4.7 (1.3)
    Walking subscale | 4.1 (1.8) | 3.7 (1.6) | 3.9 (1.7)

OUTCOME MEASURES:

1. Primary Outcome: Daily Time in Moderate/Vigorous Physical Activity
Description: Time spent in Moderate/Vigorous Physical Activity (MVPA) was measured with a SenseWear Mini sensor over a 7-day period. The mean time was calculated in bouted MVPA per day. A bout is defined as >= 10 consecutive minutes or more at the level of >= 3 METs (i.e., the lower bound of MVPA), with allowance for interruption of up to two minutes below the threshold.
Time Frame: Baseline, 9 weeks, 18 weeks, 27 weeks
Population: 59 participants were randomized into each group. Week 9: Immediate Group - 3 withdrew;1 with missing data. Delay Group - 2 withdrew Week 18: Immediate Group - 3 additional participants withdrew; 2 with missing data. Delay Group - 1 additional participant withdrew.
  Week 27: Immediate Group - 1 additional participants withdrew, Delay Group - no additional participant withdrew; 6 with missing data.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Immediate Group | Delay Group
Number analyzed (Participants) | 59 | 59
Minutes
  Baseline | 37.8 (39.6) | 31.6 (42.7)
  9 weeks: number analyzed (Participants) | 55 | 57
  9 weeks | 44.7 (41.2) | 31.6 (32.4)
  18 weeks: number analyzed (Participants) | 51 | 56
  18 weeks | 43.2 (48.2) | 32.8 (36.8)
  27 weeks: number analyzed (Participants) | 50 | 52
  27 weeks | 37.8 (38.8) | 34.0 (36.1)
Statistical Analysis 1: Comparison: Immediate Group vs Delay Group; We performed an intent-to-treat analysis. For the main comparison, we used analysis of covariance (ANCOVA) to estimate an adjusted mean difference comparing time in MVPA at 9 weeks (primary end point) between groups, adjusting for baseline MVPA, diagnosis, and blocking; Test type: Superiority; Adjusted difference in mean change = 9.4, 95% CI 2-sided [-0.5 to 19.3]

2. Secondary Outcome: Time Spent in Sedentary Activity
Description: Time spent in sedentary activity was measured with a SenseWear Mini sensor over a 7-day period. The mean daily time spent in sedentary activity was calculated with an energy expenditure of <=1.5 METs, occurring in bouts of >= 20 minutes during waking hours.
Time Frame: Baseline, 9 weeks, 18 weeks, 27 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Immediate Group | Delay Group
Number analyzed (Participants) | 59 | 59
Minutes
  Baseline | 491.6 (192.5) | 523.0 (194.4)
  9 weeks: number analyzed (Participants) | 55 | 57
  9 weeks | 508.4 (203.5) | 530.0 (180.2)
  18 weeks: number analyzed (Participants) | 51 | 56
  18 weeks | 507.8 (195.8) | 531.4 (165.4)
  27 weeks: number analyzed (Participants) | 50 | 52
  27 weeks | 506.8 (179.7) | 498.0 (155.6)
Statistical Analysis 1: Comparison: Immediate Group vs Delay Group; We performed an intent-to-treat analysis. For the main comparison, we used analysis of covariance (ANCOVA) to estimate an adjusted mean difference comparing sedentary time at 9 weeks (primary end point) between groups, adjusting for baseline sedentary time, diagnosis, and blocking; Test type: Superiority; Adjusted difference in mean change = -10.4, 95% CI 2-sided [-53.4 to 32.6]

3. Secondary Outcome: Fatigue Severity Scale
Description: The Fatigue Severity Scale consists of 9 questions and measures the impact of fatigue. A total score is calculated by averaging the rating from each question. Range 1-7; lower score = less fatigue.
Time Frame: Baseline, 9 weeks, 18 weeks, 27 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Group | Delay Group
Number analyzed (Participants) | 59 | 59
score on a scale
  Baseline | 4.8 (1.4) | 4.9 (1.3)
  9 weeks: number analyzed (Participants) | 55 | 57
  9 weeks | 4.5 (1.3) | 4.9 (1.3)
  18 weeks: number analyzed (Participants) | 51 | 56
  18 weeks | 4.8 (1.3) | 4.6 (1.5)
  27 weeks: number analyzed (Participants) | 50 | 52
  27 weeks | 4.5 (1.4) | 4.7 (1.4)
Statistical Analysis 1: Comparison: Immediate Group vs Delay Group; We performed an intent-to-treat analysis. For the main comparison, we used analysis of covariance (ANCOVA) to estimate an adjusted mean difference comparing time in the Fatigue Severity Scale at 9 weeks (primary end point) between groups, adjusting for baseline fatigue score, diagnosis, and blocking; Test type: Superiority; Adjusted difference in mean change = -0.31, 95% CI 2-sided [-0.63 to 0.01]

4. Secondary Outcome: McGill Pain Questionnaire Short Form (MPQ-SF)
Description: The MPQ-SF contains 15 pain-related words, which can be rated from 0 to 3. Range 0 - 45; higher=more severe pain.
Time Frame: Baseline, 9 weeks, 18 weeks, 27 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Group | Delay Group
Number analyzed (Participants) | 59 | 59
score on a scale
  Baseline | 13.3 (10.8) | 13.9 (9.5)
  9 weeks: number analyzed (Participants) | 55 | 57
  9 weeks | 10.9 (8.4) | 14.6 (9.7)
  18 weeks: number analyzed (Participants) | 51 | 56
  18 weeks | 10.6 (9.6) | 12.6 (10.0)
  27 weeks: number analyzed (Participants) | 50 | 52
  27 weeks | 11.8 (10.0) | 11.0 (9.8)
Statistical Analysis 1: Comparison: Immediate Group vs Delay Group; We performed an intent-to-treat analysis. For the main comparison, we used analysis of covariance (ANCOVA) to estimate an adjusted mean difference comparing pain at 9 weeks (primary end point) between groups, adjusting for pain score, diagnosis, and blocking; Test type: Superiority; Adjusted difference in mean change = -2.45, 95% CI 2-sided [-4.78 to -0.13]

5. Secondary Outcome: The Patient Health Questionnaire-9 (PHQ-9)
Description: The PHQ-9 consists of nine questions (rated from 0 to 3) that correspond to nine diagnostic criteria for major depressive disorder. Range 0-27; lower score = less depressive symptoms),
Time Frame: Baseline, 9 weeks, 18 weeks, 27 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Group | Delay Group
Number analyzed (Participants) | 59 | 59
score on a scale
  Baseline | 7.6 (5.9) | 8.1 (5.6)
  9 weeks: number analyzed (Participants) | 55 | 57
  9 weeks | 6.8 (5.6) | 7.9 (5.7)
  18 weeks: number analyzed (Participants) | 51 | 56
  18 weeks | 6.0 (5.0) | 6.2 (5.4)
  27 weeks: number analyzed (Participants) | 50 | 52
  27 weeks | 5.2 (3.8) | 6.7 (5.9)
Statistical Analysis 1: Comparison: Immediate Group vs Delay Group; We performed an intent-to-treat analysis. For the main comparison, we used analysis of covariance (ANCOVA) to estimate an adjusted mean difference comparing the PHQ-9 scores at 9 weeks (primary end point) between groups, adjusting for baseline score, diagnosis, and blocking; Test type: Superiority; Adjusted difference in mean change = -0.22, 95% CI 2-sided [-1.78 to 1.35]

6. Secondary Outcome: Partners In Health Scale
Description: The Partners in Health Scale is a 12-item measure designed to assess self-efficacy, knowledge of health conditions and treatment, and self-management behaviors such as adopting a healthy lifestyle. Range 0-96; higher score = higher perceived confidence and ability in self-care.
Time Frame: Baseline, 9 weeks, 18 weeks, 27 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Group | Delay Group
Number analyzed (Participants) | 59 | 59
score on a scale
  Baseline | 72.8 (11.7) | 73.5 (12.2)
  9 weeks | 75.5 (12.5) | 74.6 (11.2)
  18 weeks | 77.7 (11.4) | 78.7 (10.8)
  27 weeks | 77.9 (12.6) | 77.4 (10.7)
Statistical Analysis 1: Comparison: Immediate Group vs Delay Group; We performed an intent-to-treat analysis. For the main comparison, we used analysis of covariance (ANCOVA) to estimate an adjusted mean difference comparing the Partners In Health Scale scores at 9 weeks (primary end point) between groups, adjusting for baseline score, diagnosis, and blocking; Test type: Superiority; Adjusted difference in mean change = 1.58, 95% CI 2-sided [-1.02 to 4.18]

7. Secondary Outcome: The Self-Reported Habit Index (SRHI) - Sitting at Work Index
Description: The SRHI is a 12-item scale, rated on a 7-point Likert scale, that measures characteristics of habitual behavior. Participants rated their strength of habit of sitting at work. A higher score indicates a stronger habit or behavior that is done frequently, automatically, and done without thinking about it. Range 1-7; higher score = stronger habit.
Time Frame: Baseline, 9 weeks, 18 weeks, 27 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Group | Delay Group
Number analyzed (Participants) | 59 | 59
score on a scale
  Baseline | 4.5 (1.7) | 4.6 (1.8)
  9 weeks | 4.3 (1.8) | 4.7 (1.7)
  18 weeks | 4.6 (1.7) | 4.6 (1.8)
  27 weeks | 4.4 (1.4) | 4.6 (1.7)
Statistical Analysis 1: Comparison: Immediate Group vs Delay Group; We performed an intent-to-treat analysis. For the main comparison, analysis of covariance (ANCOVA) was used to estimate an adjusted mean difference comparing the Sitting at Work index scores at 9 weeks (primary end point) between groups, adjusting for baseline score, diagnosis, and blocking; Test type: Superiority; Adjusted difference in mean change = 0.05, 95% CI 2-sided [-0.05 to 0.16]

8. Secondary Outcome: The Self-Reported Habit Index (SRHI) - Sitting at Leisure Index
Description: The SRHI is a 12-item scale, rated on a 7-point Likert scale, that measures characteristics of habitual behavior. Participants rated their strength of habit of sitting at leisure. A higher score indicates a stronger habit or behavior that is done frequently, automatically, and done without thinking about it. Range 1-7; higher score = stronger habit.
Time Frame: Baseline, 9 weeks, 18 weeks, 27 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Group | Delay Group
Number analyzed (Participants) | 59 | 59
score on a scale
  Baseline | 4.7 (1.4) | 4.7 (1.3)
  9 weeks: number analyzed (Participants) | 55 | 57
  9 weeks | 4.7 (1.3) | 4.8 (1.4)
  18 weeks: number analyzed (Participants) | 51 | 56
  18 weeks | 4.6 (1.3) | 4.8 (1.2)
  27 weeks: number analyzed (Participants) | 50 | 52
  27 weeks | 4.6 (1.3) | 4.7 (1.4)
Statistical Analysis 1: Comparison: Immediate Group vs Delay Group; We performed an intent-to-treat analysis. For the main comparison, analysis of covariance (ANCOVA) was used to estimate an adjusted mean difference comparing the Sitting at Leisure index scores at 9 weeks (primary end point) between groups, adjusting for baseline score, diagnosis, and blocking; Test type: Superiority; Adjusted difference in mean change = 0, 95% CI 2-sided [-0.37 to 0.37]

9. Secondary Outcome: The Self-Reported Habit Index (SRHI) - Walking Index
Description: The SRHI is a 12-item scale, rated on a 7-point Likert scale, that measures characteristics of habitual behavior. Participants rated their strength of walking habit. A higher score indicates a stronger habit or behavior that is done frequently, automatically, and done without thinking about it. Range 1-7; higher score = stronger habit.
Time Frame: Baseline, 9 weeks, 18 weeks, 27 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Group | Delay Group
Number analyzed (Participants) | 59 | 59
score on a scale
  Baseline | 4.1 (1.8) | 3.7 (1.6)
  9 weeks: number analyzed (Participants) | 55 | 57
  9 weeks | 4.4 (1.7) | 3.6 (1.7)
  18 weeks: number analyzed (Participants) | 51 | 56
  18 weeks | 4.3 (1.6) | 4.0 (1.6)
  27 weeks: number analyzed (Participants) | 50 | 52
  27 weeks | 4.7 (1.5) | 4.0 (1.7)
Statistical Analysis 1: Comparison: Immediate Group vs Delay Group; We performed an intent-to-treat analysis. For the main comparison, analysis of covariance (ANCOVA) was used to estimate an adjusted mean difference comparing the Walking index scores at 9 weeks (primary end point) between groups, adjusting for baseline score, diagnosis, and blocking; Test type: Superiority; Adjusted difference in mean change = 0.54, 95% CI 2-sided [0.08 to 0.99]

ADVERSE EVENTS:
Time Frame: 26 weeks
Description: Self-reported adverse events were collected, including muscle pain, ligament sprain, or falls while being physically active, were collected.
Arm/Group | Immediate Group | Delay Group
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/59
Other Adverse Events (participants affected / at risk) | 13/59 | 10/59
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Immediate Group (N=59) | Delay Group (N=59)
Muscle pain (Musculoskeletal and connective tissue disorders) | 10 | 9
Ligament sprain (Musculoskeletal and connective tissue disorders) | 3 | 1

LIMITATIONS AND CAVEATS:
A limitation is the inclusion of only individuals with rheumatoid arthritis and systemic lupus erythematosus. We focused on these 2 diseases because of feasibility for recruitment in our community. The findings, however, are not generalizable to people with other types of inflammatory arthritis. Furthermore, the results may not be generalizable to men because 89% of the participants were women.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-09): https://cdn.clinicaltrials.gov/large-docs/74/NCT02554474/Prot_SAP_000.pdf